CLINICAL TRIAL: NCT00601939
Title: Group Interventions for Abused, Suicidal Black Women
Brief Title: Effectiveness of Empowerment Group Sessions for Treating Suicidal African American Women in Abusive Relationships
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Nadine Kaslow, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00045774; R01MH078002 (NIH)
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Battered Women; Suicide, Attempted
Keywords: Abused; Female; African American; Group Empowerment Psychoeducational Intervention; Enhanced Treatment as Usual
MeSH Terms: conditions — Suicide, Attempted

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psychoeducational intervention (PEI) (Experimental): Culturally competent group empowerment psychoeducational treatment (group intervention that is culturally informed and educational in nature)
  Interventions: Behavioral: Psychoeducational intervention (PEI)
- Enhanced Treatment as Usual (Active Comparator): Enhanced treatment as usual that includes an adherence protocol (regular care at the hospital plus an adherence protocol)
  Interventions: Behavioral: Enhanced treatment as usual (ETAU)

INTERVENTIONS:
Behavioral: Psychoeducational intervention (PEI) — PEI consists of 10 culturally competent group empowerment psychoeducational sessions. The sessions are directed by a treatment manual and are co-led by two therapists. The sessions are guided by the theory of triadic influence (TTI) model, which incorporates cultural-environmental influences, social-situational influences, and intrapersonal influences into treatment.
  Other Names: Theory of triadic influence
  Arms: Psychoeducational intervention (PEI)
Behavioral: Enhanced treatment as usual (ETAU) — ETAU contains an adherence protocol plus access to weekly support group and a resource room.
  Arms: Enhanced Treatment as Usual

SUMMARY:
This study will evaluate the effectiveness of culturally competent psychoeducational empowerment sessions in treating suicidal African-American women who are in abusive relationships.

DETAILED DESCRIPTION:
Most suicide attempts are a sign of great distress, often originating from depression; physical and sexual abuse; substance abuse; or family history of suicide, violence, or mental disorder. Risk factors for suicidal behavior are diverse, differing with gender, age, and ethnicity. Since the mid-1980s, the number of reported suicides and suicidal thoughts among young black individuals has increased alarmingly. The higher rates may be caused by high stress living situations attributed to poverty, abuse, discrimination, racism, and difficult family life. Therefore, cultural environments, social situations, and intrapersonal influences are important considerations in developing an effective therapy to prevent suicide. This study will evaluate the effect of culturally competent psychoeducational empowerment sessions in treating suicidal African-American women who are in abusive relationships.

The participants in this single-blind study will be randomly placed in one of two treatment groups. One group will receive psychoeducational intervention (PEI) and the other will receive enhanced treatment as usual (ETAU). After screening, eligible participants will complete a 2-hour survey about life events, concerns, and feelings with a research team member. One week later, participants will complete a second 1-hour survey. Participants will then be randomly placed in the treatment groups. Participants in both groups will receive treatment at Grady Health System, but those in the PEI group will also attend 10 weekly, 90-minute group sessions. The PEI empowerment group sessions will incorporate cultural, social, and intrapersonal elements. The ETAU group will be given mental health treatment as usual plus an adherence enhancement protocol. Follow-up surveys will occur at Week 10 (after treatment completion) and at Months 6 and 12 post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Identifies as an African-American female
* Abusive relationship within the 12 months prior to study entry
* Suicide attempt within the 12 months prior to study entry
* Seeks services at Grady Health System

Exclusion Criteria:

* Score of less than 22 on Mini Mental Status Exam (MMSE)
* Score of less than 18 on Rapid Estimate of Adult Literacy in Medicine (REALM)
* Acutely psychotic

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 397 (Estimated)
Dates: Start 2008-03; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in Beck Scale for Suicide Ideation Score | Baseline, Week 10, Post-treatment Months 6 and 12
  The Beck Scale for Suicide (BSS) Ideation consists of 19 items with responses rated on a scale from 0 to 2. Total scores range from 0 to 38 with higher scores indicating greater feelings of suicide ideation.
Change in Suicide Attempt Index | Baseline, Week 10, Post-treatment Months 6 and 12
  Created for this study, this qualitative screening measure asks if participants have engaged in the suicidal behaviors of intentionally overdosing, cutting self, tried to shoot self or jump from a high place, tried to take life, and attempting suicide.
Change in Index of Spouse Abuse Score | Baseline, Week 10, Post-treatment Months 6 and 12
  The Index of Spouse Abuse (ISA) is a 30-item instrument where participants report how frequently abuse situations occur where 1 = never and 5 = very frequently. Total scores range from 30 to 150 and higher scores indicate a higher degree of abuse.

SECONDARY OUTCOMES:
Change in Beck Depression Inventory- II | Baseline, Week 10, Post-treatment Months 6 and 12
  The Beck Depression Inventory-II is a 21-item questionnaire where items are scored from 0 to 3, with higher scores assigned to more severe symptoms. Total scores range from 0 to 63, with higher scores indicating greater severity of depressive symptoms.
Change in Beck Hopelessness Scale | Baseline, Week 10, Post-treatment Months 6 and 12
  The Beck Hopelessness Scale is a 20-item instrument where each statement is answered as being true or false. Optimistic responses are scored as 0 while pessimistic responses are scored as 1. Total scores range from 0 to 20 and higher scores indicate greater feelings of hopelessness.
Change in Self-Efficacy Scale for Battered Women | Baseline, Week 10, Post-treatment Months 6 and 12
  The Self-Efficacy Scale for Battered Women is a 12-item instrument where participants report how confident they are about performing tasks related to asking for help and taking control of their lives. Items are scored on a scale of 0 to 100 where 0 = couldn't do it at all and 100 = completely sure I could do it. Total raw scores range from 1 to 1200, where higher scores indicate increased self efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine J. Kaslow, PhD, Principal Investigator — Emory University
Locations (1):
- Grady Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617